CLINICAL TRIAL: NCT07244172
Title: Effects of Mud-walk on Foot Posture and Balance in Children With Flexible Flatfeet
Brief Title: Foot Posture and Balance in Children With Flexible Flatfeet: Effects of Mud-walk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REC/RCR&AHS/SAMANMAQBOOL
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Flexible Flatfoot
Keywords: Balance; Flexible Flatfoot; Foot Posture; Foot Posture Index; Navicular Drop Test; Pediatric Berg Balance Scale
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: This quasi-experimental study aims to determine effects of mud-walk on foot posture and balance in children with flexible flatfeet. The study will involve 37 children with bilateral flexible flatfeet of age 6-11 years. The navicular height, foot posture, balance and functional performance of lower limb will be assessed through Navicular Drop Test, Foot Posture Index-6, Pediatric Berg Balance Scale and Single Leg Hop Test respectively. All recruited children will receive intervention for 30 minutes a day for 3 days a week for total 6 weeks. The exercise program will include warm up phase, walk on mud and cool down phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mud training (Other): The children will walk on within a rectangular boundary of "2 × 8 dimension" (2 feet by 8 feet) with 5 cm depth. The exercise program will have 3 phases: warm up, walk on mud and cool down. The warm up phase will consist of stretching of the hamstring muscles using the static technique. The main exercise program will include walk on mud in four manners and progression will be added after 3 weeks.
  Interventions: Other: mud-walk

INTERVENTIONS:
Other: mud-walk — * The participants will walk on the mud within a rectangular boundary of "2 × 8 dimension" (2 feet by 8 feet) with 5 cm depth.
  * The exercise program will have 3 phases: warm up, walk on mud and cool down.
  * The warm up phase will consist of stretching of the hamstring muscles using the static technique.
  The main exercise phase will consist of 20 minutes of walk on mud in four manners with each manner for 5 minutes:
  1. forward walk
  2. back ward walk
  3. sideways walk
  4. S-shaped or figure-eight walk After 3 weeks, while walking in each manner the participants will pick up small objects (soft balls) with toes from mud and place them elsewhere.
  The cool down phase will consist of 5 minutes and will include
  * soaking feet in water
  * washing with soap
  * rinsing with clean water,
  * drying with towel
  * application of emollient

SUMMARY:
The study will be a quasi-experimental study with a pre-post study design. 37 children with bilateral flexible flatfeet of age 6-11 years will be recruited by non-probability convenience sampling with pre and post assessment. The navicular height, foot posture, balance and functional performance of lower limb will be assessed through Navicular Drop Test, Foot Posture Index-6, Pediatric Berg Balance Scale and Single Leg Hop Test respectively. All recruited children will receive intervention for 30 minutes a day for 3 days a week for total 6 weeks. The exercise program will include warm up phase, walk on mud and cool down phase. Data will be analyzed through SPSS version 27.0.

DETAILED DESCRIPTION:
Flatfeet is one of the predominant conditions of feet in children and is characterized by absence of medial longitudinal arch. Flatfeet affect the foot posture by altering the entire biomechanics of musculoskeletal system of lower limb. It ultimately affects the balance and functional mobility in children and may have poor quality of life in adulthood. The strength training programs and uneven surfaces have been used previously for its intervention. The mud-walk provides natural resistance along with sensory feedback due to its soft, variable surface. The aim of this study is to determine effects of mud-walk on foot posture, balance and functional performance of lower limb in children with flexible flatfeet.

The study will be a quasi-experimental study with a pre-post study design. 37 children with bilateral flexible flatfeet of age 6-11 years will be recruited by non-probability convenience sampling with pre and post assessment from Presentation Convent High School and The Sanai School Sargodha. All children will be assessed for inclusion and exclusion. The navicular height, foot posture, balance and functional performance of lower limb will be assessed through Navicular Drop Test, Foot Posture Index-6, Pediatric Berg Balance Scale and Single Leg Hop Test respectively. All recruited children will receive intervention for 30 minutes a day for 3 days a week for total 6 weeks. The exercise program will include warm up phase, walk on mud and cool down phase. Data will be analyzed through SPSS version 27.0.

ELIGIBILITY:
Inclusion Criteria:

* Children with bilateral flexible flat feet
* Children aged 6-11 years
* Children who are not involved in any other trial
* FPI-6 score >6

Exclusion Criteria:

* Children with rigid flatfeet
* Prior foot or ankle surgery
* Pain in lower extremities
* Overweight or obese
* Any other foot deformities
* Any neurological or neuromuscular disorder

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Foot Posture Index-6 (FPI-6) | Baseline and 6th week
  FPI-6 is a clinical tool for quantifying foot positioning that uses established criteria. The FPI consists of the following six items, each graded on a scale of -2 to +2 referring to the position of the forefoot, midfoot and hindfoot, and the three planes of motion:
  1. talar head palpation;
  2. symmetry of supra and infra lateral malleolar curvature;
  3. inversion/eversion of the calcaneus;
  4. prominence in the region of the talus-navicular joint;
  5. height of the medial longitudinal arch;
  6. abduction/adduction of the forefoot. The FPI thus obtained ranges from -12 (highly supinated) to +12 (highly pronated).
  It can be
  * highly pronated (+10 to +12)
  * pronated (+6 to +9)
  * normal (0 to +5)
  * supinated (-1 to -4)
  * highly supinated (-5 to -12). FPI-6 demonstrates a perfect weighted kappa value (Kw = 0.86), with a high intra-rater reliability (ICC = 0.96)
Navicular Drop Test (NDT) | Baseline and 6th week
  Navicular Drop Test is used to evaluate the amount of foot pronation. It is considered as a reliable and valid tool to measure static navicular height. The navicular height is measured while the child is sitting with barefoot flat on a platform with 90◦ knee flexion and the subtalar joint in neutral position. The Navicular drop is recorded as the difference in navicular height between subtalar joint neutral position and relaxed standing. Navicular drop more than 9 mm represented a pronated foot type, 5-9 mm a neutral foot and less than 5 mm a supinated foot. This test's intra-rater and inter-rater reliability has been demonstrated to range from 0.73 to 0.96 .
Pediatric Berg Balance Scale (PBBS) | Baseline and 6th week
  A 14-item criterion-referenced measure that examines functional balance in the context of everyday tasks in the pediatric population. Each item level scores range from 0-4 which is determined by the ability to perform the assessed activity. Maximum score = 56 points with 56 points being a perfect score. Test-retest (ICC2,1 = 0.923), interrater (ICC2,1 = 0.972), and intra-rater (ICC2,1 = 0.895-0.998) are reliabilities of PBS. It has high internal consistency (Cronbach α = 0.94) .

SECONDARY OUTCOMES:
Single Leg Hop Test | Baseline and 6th week
  Single leg hop test assesses functional performance of lower limb. The test method involves performing a forward jump, covering the maximum possible distance with one foot, landing on the same foot, and finally maintaining balance for at least 2 seconds. After performing 2 or 3 attempts, the individual executes a complete single-leg hop with the dominant leg, and the distance covered is recorded. An intra-class correlation coefficient (ICC) of over 0.85 has been reported for the reliability of this test in various studies.

CONTACTS AND LOCATIONS:
Overall Officials: Saman Maqbool, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Markowicz M, Skrobot W, Labuc A, Poszytek P, Orlikowska A, Perzanowska E, Krasowska K, Drewek K, Kaczor JJ. The Rehabilitation Program Improves Balance Control in Children with Excessive Body Weight and Flat Feet by Activating the Intrinsic Muscles of the Foot: A Preliminary Study. J Clin Med. 2023 May 9;12(10):3364. doi: 10.3390/jcm12103364. PMID 37240471